CLINICAL TRIAL: NCT01263431
Title: Prospective Randomized Trial on Surgical Treatment of Grade 3 Hemorrhoids: Hemorrhoidectomy Versus Doppler-guided Transanal Haemorrhoidal Dearterialisation and Anopexy
Brief Title: Comparison Between Excisional Hemorrhoidectomy and Haemorrhoidal Dearterialisation With Anopexy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Paola De Nardi, MD, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Emorroidi grado 3
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Third Degree Hemorrhoids
Keywords: Hemorrhoidectomy, haemorrhoidal dearterialisation, anopexy
MeSH Terms: interventions — Hemorrhoidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemorrhoidectomy (Active Comparator): Excision of hemorrhoid cushions
  Interventions: Procedure: Hemorrhoidectomy
- Hemorrhoidal dearterialization (Experimental): Ligation of therminbal branches oh hemorrhoid arteries
  Interventions: Procedure: Hemorrhoidal dearterialization

INTERVENTIONS:
Procedure: Hemorrhoidectomy — Each of the main haemorrhoid is dissected and the apex is ligated and then cut, near to the dentate line
  Arms: Hemorrhoidectomy
Procedure: Hemorrhoidal dearterialization — A special instrument (THD, G.F., Medical Division, Correggio, Italy )with an incorporated Doppler probe is used to detected the six terminal branches of the superior rectal artery which are ligated above the dentate line, then a running suture is performed in order to obtain a mucopexy
  Arms: Hemorrhoidal dearterialization

SUMMARY:
Aim of the study is to compare short term results of 2 surgical treatment for grade 3 hemorrhoidal disease, namely: pain and postoperative morbidity,complications and effectiveness within 30 days, re-starting daily and working activity, patients' satisfaction

DETAILED DESCRIPTION:
Excisional haemorrhoidectomy is burdened by severe postoperative pain. For this reason less painful treatments have been developed, such as Doppler-guided haemorrhoidal artery ligation and stapled anopexy. Both techniques seem to be safe, causing little postoperative pain. A combination of the two techniques could possibly treat both bleeding and prolapse with minimal discomfort

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80, candidate to surgery for 3rd degree hemorrhoids

Exclusion Criteria:

* Previous anal surgery or pelvic radiotherapy
* Fecal incontinence or obstructed defecation
* IBD, IBS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 1 week

SECONDARY OUTCOMES:
postoperative morbidity | 30 days
resumption of working activity | 30 days
patient's satisfaction | 30 days
Relapse | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Paola De Nardi, MD, Principal Investigator — San Raffaele Scientific Institute
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Derived] De Nardi P, Capretti G, Corsaro A, Staudacher C. A prospective, randomized trial comparing the short- and long-term results of doppler-guided transanal hemorrhoid dearterialization with mucopexy versus excision hemorrhoidectomy for grade III hemorrhoids. Dis Colon Rectum. 2014 Mar;57(3):348-53. doi: 10.1097/DCR.0000000000000085. PMID 24509458